CLINICAL TRIAL: NCT01845363
Title: Antibiotic Prophylaxis in Bariatric Surgery With Continuous Infusion of Cefazolin: Determination of Concentration in Adipose Tissue
Brief Title: Antibiotic Prophylaxis in Bariatric Surgery With Cefazolin: Concentration in Adipose Tissue
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Rafael Anlicoara, Master´s degree, Universidade Federal de Pernambuco
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Cefa01
Record Dates: First submitted 2013-04-29; First posted 2013-05-03 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-04

CONDITIONS: Obesity
Keywords: Obesity; Bariatric surgery; Cefazolin; antimicrobial prophylaxis; administration and dosage
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cefazolin (Other): Cefazolin used in antimicrobial prophylaxis
  Cefazolin administered a first dose of 2g in anesthetic induction, followed by continuous dosage of 1g diluted in 250mL of saline solution for two hours.
  Two samples of subcutaneous tissue were collected for analysis: the first soon after the incision, and a second before skin synthesis.
  The samples were processed by High Pressure Liquid Chromatography (HPLC).
  Interventions: Drug: Cefazolin used in antimicrobial prophylaxis

INTERVENTIONS:
Drug: Cefazolin used in antimicrobial prophylaxis — Cefazolin administered a first dose of 2g in anesthetic induction, followed by continuous dosage of 1g diluted in 250mL of saline solution for two hours.
  Two samples of subcutaneous tissue were collected for analysis: the first soon after the incision, and a second before skin synthesis.
  The samples were processed by HPLC.

SUMMARY:
Eighteen patients were given a dose of 2g Cefazolin in anesthetic induction, supplemented with 1g delivered through continuous infusion during surgery. Adipose samples, obtained at the beginning and end of surgery, were analyzed using high performance liquid chromatography.

Some published studies suggest that the dose of 2g does not supply the minimum inhibitory concentration for principal causal agents of surgical site infection.

To determine the concentration of Cefazolin in adipose tissue of patients undergoing bariatric surgery and to evaluate the relationship between concentrations obtained and body mass index (BMI).

ELIGIBILITY:
Inclusion Criteria:

* body mass index greater than 35 and less than 50kg/m2

Exclusion Criteria:

* Hypotension during surgery with use of vasoactive drugs
* renal disfunction (creatinine >1.5 mg/dL)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
dosage of Cefazolin in adipose tissue during bariatric surgery | eight months

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Anlicoara, MD, Principal Investigator — UFPE; Alvaro AB Ferraz, PhD, Study Chair — UFPE - Hospital das Clínicas; José L de Lima Filho, PhD, Study Director — Laboratory of Immunopathology Keiso Asami(LIKA) - UFPE
Locations (1):
- Universidade Federal de Pernambuco - Hospital das Clínicas, Recife, Pernambuco, Brazil